CLINICAL TRIAL: NCT03563469
Title: Assessment of Salivary Bacterial Level and Dental Caries Experience in a Group of Egyptian Children With Black Stained Teeth: A Cross Sectional Study
Brief Title: Assessment of Salivary Bacterial Level and Dental Caries Experience in a Group of Egyptian Children With Black Stained Teeth
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Joanna Nassef William Samuel, master student in Cairo University, Cairo University
Other Study IDs: CEBD-CU-2015-02-26
Record Dates: First submitted 2018-06-09; First posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Black Stain Dental, Dental Black Stain, Black Stain*, Black Stains, Tooth Stains

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Salivary bacterial and pH level — 1. Saliva sample will be collection ask the patient to stop eating and drinking for one hour before collecting the sample,(2) Give the patient distilled water and ask them to rinse their mouth well for 1 min,five minutes after this oral rinse, ask the patient to spit into 50ml sterile tube, collect 5ml of saliva and return to the laboratory within an hour.
  2. The dental caries of all patients will also be recorded using dental mirror and explorer. The caries experience will be recorded in diagnostic chart using the World Health Organization (WHO) criteria for deciduous teeth and dmft caries index.
  Other Names: Dental caries experience using dmft caries index

SUMMARY:
Black stains (BS) are type of extrinsic discoloration of the tooth. It's characterized as dark lines or an incomplete coalescence of dark dots found mostly on cervical third of the crown. Most studies worldwide found that children with the black stained teeth have low caries prevalence. A study on Brazilian population also suggested that black stains might be protective factor against development of dental caries. A study reported that chromogenic bacteria were proposed as etiological factor in production of black stains.The most common microbiological composition of BS was found to be Actinomycetes. Dental examination and saliva samples collection will be done for black stained teeth children of outpatient clinic of Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University. This research adopts null hypothesis; it assumes that there is no effect on dental caries experience in children with black stained teeth.

ELIGIBILITY:
Inclusion Criteria:

* Patients with black stained teeth who were reported to outpatient clinic of Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University ranging in age between 4-6 years.
* With primary dentition.
* Both sexes will be included.
* Cooperative children.

Exclusion Criteria:

* Having oral disease (such as peridotites, salivary gland disorder, and oral mucosal disease).
* Having autoimmune disease.
* Receiving any antibiotic treatment in the past three months.
* Parents refuse to sign the consent

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Egyptian children 4-6 years old with black stained teeth.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Salivary bacterial level | 6 months
  salivary sample collection by passive drooling

SECONDARY OUTCOMES:
Dental caries experience | 6 months
  The dental caries of all patients will also be recorded using dental mirror and explorer. The caries experience will be recorded in diagnostic chart using the World Health Organization (WHO) criteria for deciduous teeth and dmft caries index
Salivary pH level | 6 months
  salivary sample collection and measured by the pH meter